CLINICAL TRIAL: NCT03229434
Title: Effects of Mountain Hiking on Physiological and Psychological Health Parameters With Special Focus on the Influence of the Environment
Brief Title: Mountain Hiking & Environmental Influences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Martin Burtscher, Prof., Universitaet Innsbruck
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ARMH_2
Record Dates: First submitted 2017-07-19; First posted 2017-07-25 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Healthy Participants
Keywords: affective responses; stress-related parameters; green exercise
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: pseudonymes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Widely pristine area (Experimental): Outdoor mountain hiking (approximately 6 hours, 8km, 800 altitude meters, estimated speed: 4km/h [uphill], 5.2km/h [downhill]) in a widely pristine area with moderate intensity (Rating of perceived exertion: ~ 11-15).
  Interventions: Behavioral: Mountain hiking
- Anthropogenically influenced area (Active Comparator): Outdoor mountain hiking (approximately 6 hours, 8km, 800 altitude meters, estimated speed: 4km/h [uphill], 5.2km/h [downhill]) in an anthropogenically influenced area with moderate intensity (Rating of perceived exertion: ~ 11-15).
  All characteristics of the hiking (duration, time, difference in altitude, ...) are planned to be comparable to the experimental condition except the area.
  Interventions: Behavioral: Mountain hiking

INTERVENTIONS:
Behavioral: Mountain hiking — Compare arm description
  Other Names: Walking

SUMMARY:
In a randomized crossover design, approximately 50 healthy participants will be randomly exposed to outdoor mountain hiking (approximately 6 hours each) in two different areas: an anthropogenically influenced area and in a widely pristine area.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation

Exclusion Criteria:

* pregnancy
* breastfeeding
* chronic or acute diseases (already existing or diagnosed during the study)
* unable to be physically active assessed by the Physical Activity Readiness Questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-29 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Cortisol (Saliva Sampling) at 6 hours | 6 hours
  Physiological response
Change from baseline subscales of mood survey scale at 6 hours | 6 hours
  Psychological response

SECONDARY OUTCOMES:
Change from baseline blood pressure at 6 hours | 6 hours
Change from baseline lung function at 6 hours | 6 hours
Change from baseline respiratory gas analysis at 6 hours | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport Science, Medical Section, University of Innsbruck, Innsbruck, Austria

REFERENCES:
- [Background] Niedermeier M, Einwanger J, Hartl A, Kopp M. Affective responses in mountain hiking-A randomized crossover trial focusing on differences between indoor and outdoor activity. PLoS One. 2017 May 16;12(5):e0177719. doi: 10.1371/journal.pone.0177719. eCollection 2017. PMID 28520774